CLINICAL TRIAL: NCT06885762
Title: Safety and Efficacy of Efgartigimod in Guillain-Barré Syndrome
Brief Title: Efgartigimod for the Treatment of Guillain-Barré Syndrome
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zhongming Qiu (Other)
Responsible Party: Sponsor-Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Organization: Xinqiao Hospital of Chongqing (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-010-01
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Guillain-Barre Syndrome (GBS)
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: efgartigimod

INTERVENTIONS:
Drug: efgartigimod — efgartigimod 20 mg/kg was administered via intravenous infusion on day 1 and day 5 of the treatment period only.

SUMMARY:
The goal of this clinical trial is to evaluating the efficacy and safety of efgartigimod in the treatment of Guillain-Barré Syndrome and exploring the immunological mechanisms of efgartigimod therapy in Guillain-Barré Syndrome. The main questions it aims to answer are:

Will efgartigimod improve the symptoms of participants? What medical problems do participants have when using efgartigimod?

Participants will:

On day 1 and day 5 of the treatment period, drug A was administered intravenously.

Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older;
2. Meet the diagnostic criteria as specified in the *European Guidelines for the Diagnosis and Treatment of Guillain-Barré Syndrome 2023 Edition*;
3. Onset of GBS symptoms within 2 weeks prior to enrollment;
4. GBS-DS score of 3-5;
5. Written informed consent obtained.

Exclusion Criteria:

1. Patients with GBS symptoms for more than 2 weeks;
2. Known hypersensitivity of the study subject to any component of the investigational drug or any other anti-neonatal Fc receptor (FcRn) agent;
3. Any uncontrolled active infection or severe infection within 8 weeks prior to screening;
4. Patients with other autoimmune diseases, such as Sjögren's syndrome, systemic lupus erythematosus, neuromyelitis optica, myasthenia gravis, multiple sclerosis, etc., requiring treatment with immunosuppressive agents;
5. Vaccination within 4 weeks prior to screening or planned vaccination during the study period;
6. Pregnant or breastfeeding, or planning to become pregnant during the study period, or women of childbearing potential not using effective contraception;
7. Currently participating in another clinical trial of similar investigational agents (FcRn antagonists);
8. Use of the investigational drug within 3 months prior to screening or within five half-lives of the drug (whichever is longer);
9. Patients with a history of malignancy, including malignant thymoma, myeloproliferative or lymphoproliferative disorders, unless considered cured by adequate treatment and without evidence of recurrence for ≥3 years prior to screening. Patients with completely resected non-melanoma skin cancer (e.g., basal cell carcinoma or squamous cell carcinoma) or carcinoma in situ of the cervix are eligible at any time;
10. Patients with clinical evidence of other significant severe diseases or who have recently undergone major surgery, which may confound study results or place the patient at undue risk. Patients with severe renal/hepatic impairment may be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-13 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Guillain-Barré Syndrome Disability Scale (GBS-DS) | 12 weeks.
  The mean time to first achieve a GBS-DS score of ≤1 within 12 weeks.